CLINICAL TRIAL: NCT03309930
Title: Narrative Comprehension by People With Acquired Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miami University (Other)
Collaborators: Duquesne University (Other); University of Nebraska Lincoln (Other); University of Arizona (Other)
Responsible Party: Principal Investigator, Kelly Knollman-Porter, Assistant Professor, Miami University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: #01377r
Record Dates: First submitted 2017-10-09; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Aphasia; Traumatic Brain Injury
Keywords: comprehension; Strategies; repeated exposure
MeSH Terms: conditions — Aphasia; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: During Study 1 participants will be exposed to three different conditions: (a) written text only, (b) auditory synthetic speech output only and (c) a combined condition (written and auditory output). During Study 2 participants will be provided repeated exposure to synthetic speech. Participants can participate in 1 or both studies with 1 study results not being dependent on the other study. .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comprehension Acquired Brain Injury (Experimental): All participants will be exposed to 3 conditions: (a) written text, (b) auditory output (synthetic speech), and combined conditions for study 1. For study 2 participants will be repeatedly exposed to synthetic speech output to determine the influence on comprehension. Participants are not required to participate in both studies.
  Interventions: Behavioral: Comprehension Acquired Brain Injury

INTERVENTIONS:
Behavioral: Comprehension Acquired Brain Injury — For study 1 participants will be exposed to 3 conditions as stated in previous descriptions and will last 1 to 2 sessions. Study 2 will begin with 1 session with the researcher lasting about 30 minutes. Then participants will be asked to complete practice at home for about 15 minutes each day for 2 weeks using a computer/iPad. Study 2 Post Testing and Maintenance Sessions 1 and 2: approximately 60 minutes per session.

SUMMARY:
The purpose of this two phase study is to evaluate comprehension by people with acquired brain injury. The phase 1 portion of the study will examine comprehension of narrative paragraphs under 3 conditions: (a) written text only, (b) auditory output only (i.e., synthetic speech - David voice) or combined written text and auditory output. The phase 2 portion of the study is to evaluate comprehension of sentences and paragraphs produced with computer generated (synthesized) speech and digitized natural speech after multiple exposures.

DETAILED DESCRIPTION:
Part 1 Experimental Procedures: Written or Spoken Paragraph Level Measure o Participants will read or listen to 12 paragraph length narrative stories in the following 3 conditions: (a) written text only, (b) auditory output only (i.e., synthetic speech - David), or combined written text and auditory output. Participants will answer 10 questions regarding the information contained in each of the 12 stories. Anticipated time requirements: 1 to 2 sessions lasting about 60 minutes each.

Part 2 Experimental Procedures: Repeated Exposures

* Independent Training Session Practice

  * To prepare the participants for independent practice (exposure) to the Synthetic 1 Condition during home training, the researchers will complete the first Independent Training Session with the participant within the clinic environment to verify participants understanding of the experimental procedure.
  * The researchers will provide written instructions with simplified language and picture support to remind the participant of the practice instructions.
  * Independent training sessions will utilize the Test of Silent Reading Efficiency and Comprehension (TOSREC) sentences recorded using the Synthetic 1 Voice Condition and the Digitized Voice Condition. TOSREC sentences are simple sentences presented at 1st, 2nd, and 3rd grade levels. Example sentence include: "A cow is an animal", and "Bears go to school". The participants will respond "yes" or "no" to each of 30 TOSREC sentences presented in a systematically randomized order. "Yes" and "no" responses will be recorded using active areas on the iPad created using a computer program designed for delivering stimuli (e.g., Blackboard, Canvas). All practice will be completed via the computer platform (e.g., Blackboard, Canvas) on the iPad. All 30 practice items should be completed in one sitting; however, the participant can take a break 5-10 minutes break during practice if needed.
  * During this first Independent Training Session Practice, the researcher will provide the participant with verbal and written instructions regarding how to access each item and ensure that the participant understands the task prior to independent practice.
* Independent Training Sessions

  * Participants will be given an iPad with Wi-Fi capabilities to use in their home (as well as a charger. Alternatively, participants may choose to use their own iPad.
  * The researchers will instruct each participant to listen to and/or reading 15 sentences per day per condition (Synthetic 1 and Digitized Sentence presentations). The researchers will provide written instructions with simplified language and picture support to remind the participant of the practice instructions.
  * The participants will respond "yes" or "no" to each of the 30 TOSREC sentences presented in a systematic randomized order. All 30 practice items should be completed in one sitting; however, the participant can take a 5-10 minute preach during practice if needed.
  * Participants will receive feedback about overall percentage performance accuracy at the end of each daily session.
  * All practice will be completed via the computer platform (e.g., Blackboard, CANVAS) on the iPad. Participants will practice for a period of two weeks (12 sessions). This is expected to take the participants no more than 15 minutes per day. The person will be asked to complete the practice up to 6 days per week. The participant will decide the days and times of practice as fits his or her schedule.

Post-Testing Sessions

* One Post-Testing Session will occur within 1 week after the last practice session ends. It will last about 60 minutes. Post-Testing tasks include responding to 45 yes/no TOSREC sentences (15 per 3 conditions), selecting a picture following the 45 Norman Rockwell sentence level comprehension task (15 per 3 conditions), and answering questions after listening to two QRI stories from one condition (Synthetic 1).

  o Following completion of the procedure above, participants will rate the accuracy and ease of comprehension of the sentences from each condition using a 5-point Likert scale. These questions appear in Appendix G.
* The Maintenance Session will occur about 4 weeks after the last practice session ends. It will last approximately 60 minutes. The Maintenance Session tasks include responding to 45 yes/no TOSREC sentences (15 per 3 conditions), selecting a picture following the Norman Rockwell sentence level comprehension task (15 per 3 conditions), and answering questions after listening to two QI stories from one condition (Synthetic 1).

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of an acquired cognitive-communication impairment secondary to brain injury/stroke
* be 19-85 years of age
* be a least, 3 months post acquired brain injury
* primarily be a speaker of American English

Exclusion Criteria:

* exhibit the presence of a hearing impairment (i.e., prescribed hearing aid or failed hearing screening)
* demonstrate a vision or motor impairment that negatively influences study completion
* Study 2: have not access to wireless internet
* Study 2: exhibit and inability to independently (or with caregiver support) use the iPad device to complete the experimental tasks.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2018-10-06 (Estimated); Study Completion 2018-10-06 (Estimated)

PRIMARY OUTCOMES:
Comprehension Across Conditions (Study 1 of 2) | Comprehension accuracy across conditions will be assessed over 1 to 2 days.
  Participants will answer 10 multiple choice questions regarding the information contained in each of the 12 stories presented in 3 conditions: (1) written text only (b) auditory output only and (c) combined written text and auditory output .
Repeated Exposure to Digitized and Synthetic Speech (Study 2 of 2) | 2 weeks
  Participants will answer 30 yes/no questions per session. Comprehension percentage accuracy will be measured over the course of 2 weeks

SECONDARY OUTCOMES:
Comprehension Generalization | measured 1 week and 4 weeks post termination of treatment
  Participants will listen to two stories presented in synthetic, computer generated speech and answer comprehension questions about the content of the stories to determine auditory comprehension accuracy
Perceived Comprehension Accuracy | measured 1 week and 4 weeks post termination of treatment
  Participants will rate the accuracy and ease of comprehension of the sentences from each condition using a 5 point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Knollman-Porter, PhD, Principal Investigator — Miami University; Sarah Wallace, PhD, Principal Investigator — Duquesne University
Locations (1):
- Miami University, Oxford, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing the data because of possible breach of privacy given the small number of local people with acquired brain injury/stroke.

REFERENCES:
- [Background] Wagner R. K., Torgesen J. K., Rashotte C. A., Pearson N. A. (2010). Test of Silent Reading Efficiency and Comprehension (TOSREC) examiner's manual. Austin, TX: Pro-Ed.